CLINICAL TRIAL: NCT01451463
Title: Impact of Xenazine(Tetrabenazine)on Gait and Functional Activity in Individuals With Huntington's Disease
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Lundbeck LLC (Industry)
Responsible Party: Principal Investigator, Sandra Kostyk, Clinical Assistant Proffessor, Ohio State University
Other Study IDs: 2010H0312
Record Dates: First submitted 2011-10-10; First posted 2011-10-13 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; Chorea; Gait; Balance
MeSH Terms: conditions — Huntington Disease; Chorea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In individuals with Huntington's disease (HD), chorea may contribute to balance problems and difficulties with walking, sit to stand transfers and stair climbing that in turn may contribute to high fall rates. Xenazine (tetrabenazine) is a monoamine-depleting drug that is commonly used to reduce chorea.

The purpose of this study is to compare: 1) spatial and temporal gait measures, 2) performance on functional mobility measures, and 3) amount of daily walking activity before and after administration of Xenazine in individuals with HD. It is hypothesized that the use of Xenazine to decrease chorea will improve functions of 1) gait, 2) sit-to-stand transfers 3) stair climbing and 4) overall daily physical activity and function.

DETAILED DESCRIPTION:
Individuals with HD who are ambulatory and are either already taking Xenazine or have been newly prescribed the medication will be recruited for this prospective open-label study. A variety of motor assessments will be preformed while subject are taking Xenazine or after a period off of the medications. These tests include: Unified Huntington's Disease Rating Scale (UHDRS) motor section, GAITRite forward walking, Tinetti Mobility Test, Timed Sit-to-Stand Test, Timed Stair Climb Test, Rhomberg test. A subset of subjects will wear an activity monitoring device on the wrist of the non-dominant hand for 5 consecutive days and nights.

ELIGIBILITY:
Inclusion Criteria:

* Huntington's Disease
* Able to ambulate independently

Exclusion Criteria:

* Other orthopedic or neurological disorder that affects gait or balance
* Pregnancy
* Chorea score <10 prior to initiation of medication.
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Huntington's disease who are already on Xenzaine (tetrabenazine) or who have recently been prescribed the medicaion.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Kostyk, MD,PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Individuals on Stable Doses of Tetrabenazine: Individuals on stable doses of tetrabenazine were studied while off medication and then following resumption of medication.
Period: Overall Study
Arm/Group | Individuals on Stable Doses of Tetrabenazine
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Individuals on Stable Doses of Tetrabenazine: 11 Individuals on stable doses of tetrabenazine were studied while off medication and then following resumption of medication.
Arm/Group | Individuals on Stable Doses of Tetrabenazine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Tinetti Mobility Test Score
Description: The Tinetti Mobility Test is a clinical test used to assess balance and gait. The Balance sub-score ranges from 0-16 (with 16 reflecting better balance) while the Gait sub-score ranges from 0-12 (with 12 reflecting better gait parameters). The Total Tinetti Mobility Test Score (TMT) is a sum of the two sub-scores with a maximum score of 28. The higher the score the better the gait and balance performance. A comparison of scores off regular stable dose of tetrabenazine for >18 hours with the performance two hours after resuming tetrabenazine was made.
Time Frame: >18 hours off Stable Dose of Tetrabenazine and at 2 hours after resumption of Tetrabenazine
Measure: Mean (Standard Deviation); unit: Total Tinetti Mobility Test Score (TMT)
Groups:
- Individuals 2 Hours After Resuming Tetrabenazine: 11 Individuals on stable doses of tetrabenazine were studied on the Tinetti Mobility Test following resumption of medication > 18 hours after being off their regular stable dose of medication.
- Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr: 11 Individuals on stable doses of tetrabenazine were studied on the Tinetti Mobility Test after being off their stable dose of medication for > 18 hours
Arm/Group | Individuals 2 Hours After Resuming Tetrabenazine | Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr
Number analyzed (Participants) | 11 | 11
Total Tinetti Mobility Test Score (TMT) | 19.91 (3.53) | 17.09 (4.04)

2. Secondary Outcome: Five Times Sit to Stand Test
Description: Subjects are asked to sit in a chair with their arms across their chests and asked to stand and sit five times in a row. The time it takes to complete 5 sit to stand cycles is timed with a stop watch. Comparison is made when off stable dose of tetrabenazine for >18 hours to performance 2 hours after resumption of tetrabenazine. Lower time scores are associated with better balance.
Time Frame: >18 hours off Stable Dose of Tetrabenazine and at 2 hours after resumption of Tetrabenazine
Measure: Mean (Standard Deviation); unit: seconds to complete 5 sit to stand cycle
Groups:
- Individuals 2 Hours After Resuming Tetrabenazine: 11 Individuals on stable doses of tetrabenazine were studied on the 5 times sit to stand test following resumption of medication . > 18 hours after being off their medication.
- Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr: 11 Individuals on stable doses of tetrabenazine were studied on the 5 times sit to stand test while off medication
Arm/Group | Individuals 2 Hours After Resuming Tetrabenazine | Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr
Number analyzed (Participants) | 11 | 11
seconds to complete 5 sit to stand cycle | 12.61 (3.00) | 15.52 (3.81)
Statistical Analysis 1: Comparison: Individuals 2 Hours After Resuming Tetrabenazine vs Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr; Test type: Superiority or Other; p = .009, t-test, 2 sided

3. Other Pre Specified Outcome: Six Condition Romberg Test
Description: The Six Condition Romberg Test is used assess static balance. Subjects are tested standing with their arms crossed over their chests and are assessed for 30 seconds in the following 6 conditions: 1) feet together, 2) feet together eyes closed, 3) feet aligned in tandem heel-to-toe position eyes open, 4) feet aligned in tandem heel-to-toe position eyes closed, 5) standing in tandem position while counting backwards by 3's from 100 with eyes open, 6) standing in tandem position while counting backwards by 3's from 100 with eyes closed. Comparison of performances were made when off stable dose of tetrabenazine for > 18 hours to performance 2 hours after resumption of tetrabenazine. If a participant could not hold a stance for the full 30 seconds, then that component of the Romberg test ended at that point with the time of that component scored in seconds; 30 seconds being the maximum score for each of the 6 tests. The total score was calculated as a sum of all of the 6 subset scores.
Time Frame: >18 hours off Stable Dose of Tetrabenazine and at 2 hours after resumption of Tetrabenazine
Measure: Mean (Standard Deviation); unit: Six Condition Romberg Test score
Groups:
- Individuals Resuming Their Stable Doses of Tetrabenazine: 11 Individuals on stable doses of tetrabenazine were studied two hours after resuming their medication after being off medication for > 18 hours.
- Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr: 11 Individuals who have been on stable doses of tetrabenazine were studied after being off medication for > 18 hours.
Arm/Group | Individuals Resuming Their Stable Doses of Tetrabenazine | Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr
Number analyzed (Participants) | 11 | 11
Six Condition Romberg Test score | 83.08 (27.57) | 73.26 (16.29)
Statistical Analysis 1: Comparison: Individuals Resuming Their Stable Doses of Tetrabenazine vs Individuals Off Their Stable Dose of Tetrabenazine for > 18 hr; Test type: Superiority or Other; p = .114, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Individuals on Stable Doses of Tetrabenazine
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No